CLINICAL TRIAL: NCT00253370
Title: A Phase II Study to Evaluate Overall Response Rate of BAY 43-9006 (Sorafenib) Combined With Docetaxel and Cisplatin or Oxaliplatin in the Treatment of Metastatic or Advanced Unresectable Gastric and Gastroesophageal Junction (GEJ) Adenocarcinoma
Brief Title: Sorafenib, Docetaxel, and Cisplatin in Treating Patients With Metastatic or Advanced Gastric or Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02951; NCI-2012-02951 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E5203 (Other: Eastern Cooperative Oncology Group (ECOG)); U10CA021115 (NIH)
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2013-12

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Metastatic Gastric Cancer; Advanced Unresectable Gastric Cancer
Keywords: Sorafenib; Docetaxel; Cisplatin; gastric cancer; gastroesophageal junction adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — Sorafenib; Docetaxel; Cisplatin; Platinum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BAY 43-9006, docetaxel, cisplatin (Experimental): Patients receive oral BAY 43-9006 400mg twice daily on days 1-21. Patients also receive docetaxel IV, 75 mg/m2 over 1 hour and cisplatin IV, 75 mg/m2 over 1-2 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: BAY 43-9006; Drug: docetaxel; Drug: cisplatin

INTERVENTIONS:
Drug: BAY 43-9006 — Given orally
  Other Names: Sorafenib (NSC724772); BAY 54-9085 (tosylate salt)
Drug: docetaxel — Given IV
  Other Names: Taxotere; RP 56976; NSC #628503
Drug: cisplatin — Given IV
  Other Names: Cis-diaminedichloroplatinum; Cis-diaminedichloroplatinum (II); diaminedichloroplatinum; cis-platinum; platinum; Platinol; Platinol-AQ; DDP; CDDP; DACP; NSC 119875.

SUMMARY:
This phase II trial is studying how well giving sorafenib together with docetaxel and cisplatin works in treating patients with metastatic or locally advanced gastric or gastroesophageal junction cancer that cannot be removed by surgery. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as docetaxel and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving sorafenib together with docetaxel and cisplatin may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the response rate (complete response and partial response) of the combination of BAY 43-9006 with docetaxel and cisplatin or oxaliplatin in patients with gastric and GEJ adenocarcinoma.

II. To evaluate the progression-free survival (PFS) and overall survival.

III. To evaluate the toxicities of BAY 43-9006 in patients with advanced and metastatic gastric or GEJ adenocarcinoma combined with docetaxel/cisplatin or docetaxel/oxaliplatin.

IV. To evaluate Raf status in the tumor and to correlate response and PFS to the presence or absence of an activating mutation in B-Raf.

V. To analyze the pharmacokinetic and pharmacogenetic properties of BAY 43-9006 including angiogenesis, monooxygenases, polymorphisms and multidrug-resistance (MDR). This study will be conducted via the E1Y03 mechanism.

OUTLINE: This is an open-label, multicenter study. Patients are stratified according to Siewert's tumor location (I vs II vs III) and extent of disease (locally advanced unresectable vs distant metastases).

Patients receive oral BAY 43-9006 twice daily on days 1-21. Patients also receive docetaxel intravenously (IV) over 1 hour and cisplatin IV over 1-2 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 3 years.

An addition of an arm containing oxaliplatin was proposed after meeting the accrual goal but did not move forward and the study was closed to accrual in July, 2007 with a final accrual of 44 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have measurable, histologically confirmed, advanced unresectable or metastatic gastric or GEJ adenocarcinoma; imaging studies must be conducted within 4 weeks of study entry
* For patients with GEJ adenocarcinoma, the tumor location should be specified using the Siewert classification used in other NCI-sponsored Phase II studies in these disease sites
* Patients must have an ECOG performance status of 0-1
* Patients may have had adjuvant chemotherapy or chemoradiation therapy, with or without 5-Fluorouracil if the treatment was performed more than 6 months before any evidence of recurrent or metastatic disease
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Must have the following baseline laboratory values obtained within 2 weeks of registration:

  * Absolute Granulocyte Count >= 1,500/mm^3
  * Platelet Count >= 100,000/mm^3
  * White Blood Count >= 3,000/mm^3
  * Serum Creatinine <= 1.5 mg/dl
  * Total Bilirubin <= 2.0 mg/dl
  * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT)/alkaline phosphatase (Alk phos) <= 2.5 x upper limit of normal
* Patients must be able to take oral medication without crushing, dissolving or chewing tablets

Exclusion Criteria:

* Prior radiotherapy, chemotherapy or investigational therapies, particularly inhibitors of tyrosine Kinases, signal transduction or angiogenesis in the treatment for their recurrent and/or metastatic gastric or GEJ adenocarcinoma
* Receiving any other investigational agents
* Being pregnant or breast-feeding; all females of childbearing potential must have a blood or urine test within 2 weeks prior to registration to rule out pregnancy
* HIV-positive patients receiving combination antiretroviral therapy are excluded from the study because of possible pharmacokinetic interactions with BAY 43-9006
* Brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to BAY 43-9006
* Acute active infection with significant clinical intervention per physician's discretion
* Previous or concurrent malignancies are not allowed, except:

  * Non-melanoma skin cancer and in situ cervical cancer
  * Treated cancer from which the patient has been continuously disease-free for more than five years
* Other uncontrolled intercurrent illnesses including, but not limited to: uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/addictive disorders that would limit compliance with study requirements
* Evidence of bleeding diathesis
* Concurrent cytochrome P450 enzyme-inducing anti-epileptic drugs:

  * Phenytoin
  * Carbamazepine
  * Phenobarbital
  * Rifampin
  * St. John's Wort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2005-10; Primary Completion 2008-05 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Weijing Sun, MD, Study Chair — University of Pennsylvania
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States

REFERENCES:
- [Result] Sun W, Powell M, O'Dwyer PJ, Catalano P, Ansari RH, Benson AB 3rd. Phase II study of sorafenib in combination with docetaxel and cisplatin in the treatment of metastatic or advanced gastric and gastroesophageal junction adenocarcinoma: ECOG 5203. J Clin Oncol. 2010 Jun 20;28(18):2947-51. doi: 10.1200/JCO.2009.27.7988. Epub 2010 May 10. PMID 20458043

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from ECOG member institutions between October 28, 2005 and July 2, 2007. The final accrual was 44 patients.
Groups:
- BAY 43-9006, Docetaxel, Cisplatin: Patients receive oral BAY 43-9006 400 mg twice daily on days 1-21. Patients also receive docetaxel IV, 75mg/m2 over 1 hour and cisplatin IV, 75 mg/m2 over 1-2 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  BAY 43-9006: Given orally
  docetaxel: Given IV
  cisplatin: Given IV
Period: Overall Study
Arm/Group | BAY 43-9006, Docetaxel, Cisplatin
Started | 44
Completed | 1
Not Completed | 43
Not completed — Adverse Event | 18
Not completed — Disease progression | 13
Not completed — Death | 2
Not completed — Withdrawal by Subject | 6
Not completed — Non-protocol therapy | 1
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 1
Not completed — Abdominal pain due to disease | 1

BASELINE CHARACTERISTICS:
Population: All 44 patients started treatment and were considered eligible and hence were included in the analysis.
Groups:
- BAY 43-9006, Docetaxel, Cisplatin: Patients receive oral BAY 43-9006 twice daily on days 1-21. Patients also receive docetaxel IV over 1 hour and cisplatin IV over 1-2 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  BAY 43-9006: Given orally
  docetaxel: Given IV
  cisplatin: Given IV
Arm/Group | BAY 43-9006, Docetaxel, Cisplatin
Number analyzed (Participants) | 44
Age, Continuous [Median (Full Range); unit: years] | 58.4 [28.4 to 85.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 37
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients With Objective Response (Complete Response or Partial Response)
Description: Response was evaluated using RECIST (Response Evaluation Criteria in Solid Tumors) 1.0 criteria. Per RECIST criteria, complete response (CR) = disappearance of all target and non-target lesions. Partial response (PR)= >=30% decrease in the sum of the longest diameters of target lesions from baseline, and persistence of one or more non-target lesion(s) and/or the maintenance of tumor marker level above the normal limits. Objective response = CR + PR.
Time Frame: Assessed every 6 weeks until disease progression or up to 3 years
Population: All enrolled patients started treatment and were considered eligible and hence were all included in the analysis.
Measure: Number (90% Confidence Interval); unit: Proportion of patients
Groups:
- BAY 43-9006, Docetaxel, Cisplatin: Patients receive oral BAY 43-9006 twice daily on days 1-21. Patients also receive docetaxel IV, 75 mg/m2 over 1 hour and cisplatin IV, 75 mg/m2 over 1-2 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  BAY 43-9006: Given orally
  docetaxel: Given IV
  cisplatin: Given IV
Arm/Group | BAY 43-9006, Docetaxel, Cisplatin
Number analyzed (Participants) | 44
Proportion of patients | 0.409 [0.284 to 0.544]
Statistical Analysis 1: Comparison: BAY 43-9006, Docetaxel, Cisplatin; The study was designed to distinguish a response rate of 40% from 20%, the null hypothesis. With the planned sample size of 36 eligible patients, the study has 91% power based on a 0.09 level one-sided test; Test type: Superiority or Other; p = 0.0012, one-sample binomial test; proportion of participants = 0.409, 90% CI 2-sided [0.284 to 0.544]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival was defined as the shorter of:
  1. The time from registration to progression. or
  2. The time from registration to death without documentation of progression given that the death occurs within 4 months of the last disease assessment without progression (or registration, whichever is more recent).
  Therefore, cases not meeting either of the criteria for a PFS event are censored at the date of last disease assessment without progression (or registration, whichever is more recent).
  Progression is defined as at least 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s) or unequivocal progression of existing non-target lesions.
Time Frame: Assessed every 6 weeks until disease progression or up to 3 years
Population: All enrolled patients started treatment and were considered eligible and hence were all included in the analysis.
Measure: Median (90% Confidence Interval); unit: Months
Groups:
- BAY 43-9006, Docetaxel, Cisplatin: Patients receive oral BAY 43-9006 twice daily on days 1-21. Patients also receive docetaxel IV, 75 mg/m2over 1 hour and cisplatin IV, 75 mg/m2 over 1-2 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  BAY 43-9006: Given orally
  docetaxel: Given IV
  cisplatin: Given IV
Arm/Group | BAY 43-9006, Docetaxel, Cisplatin
Number analyzed (Participants) | 44
Months | 5.8 [5.4 to 7.4]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from registration to death from any cause.
Time Frame: Assessed every 3 months if patient is < 2 years from study entry; then every 6 months if patient is 2-3 years from study entry.
Population: All enrolled patients started treatment and were considered eligible and hence were all included in the analysis.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | BAY 43-9006, Docetaxel, Cisplatin
Number analyzed (Participants) | 44
Months | 13.6 [8.6 to 16.1]

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment
Arm/Group | BAY 43-9006, Docetaxel, Cisplatin
Serious Adverse Events (participants affected / at risk) | 40/44
Other Adverse Events (participants affected / at risk) | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BAY 43-9006, Docetaxel, Cisplatin (N=44)
Allergic reaction (Immune system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Leukocytes decreased (Investigations) | 18
Lymphopenia (Investigations) | 2
Neutrophils decreased (Investigations) | 28
Platelets decreased (Investigations) | 2
Atrial fibrillation (Cardiac disorders) | 1
Hypotension (Vascular disorders) | 2
Fatigue (General disorders) | 7
Weight loss (Investigations) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 10
Anorexia (Metabolism and nutrition disorders) | 6
Constipation (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 9
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 6
Fistula, Rectum (Gastrointestinal disorders) | 1
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Stenosis (incl anastomotic) esophagus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Esophagus, hemorrhage (Gastrointestinal disorders) | 1
Hemorrhage-other (Vascular disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Infection w/ gr3-4 neut, catheter relate (Infections and infestations) | 2
Infection w/ gr3-4 neut, urinary tract (Infections and infestations) | 2
Infection Gr0-2 neut, foreign body (Infections and infestations) | 1
Infection w/ gr3-4 neut, blood (Infections and infestations) | 2
Infection Gr0-2 neut, blood (Infections and infestations) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Alkaline phosphatase increased (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2
Creatinine increased (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 5
Ataxia (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Neuropathy-sensory (Nervous system disorders) | 4
Seizure (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 3
Back, pain (Musculoskeletal and connective tissue disorders) | 1
Esophagus, pain (Gastrointestinal disorders) | 1
Head/headache (Nervous system disorders) | 1
Scalp, pain (Skin and subcutaneous tissue disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BAY 43-9006, Docetaxel, Cisplatin (N=44)
Anemia (Blood and lymphatic system disorders) | 33
Leukocytes decreased (Investigations) | 19
Lymphopenia (Investigations) | 3
Neutrophils decreased (Investigations) | 16
Platelets decreased (Investigations) | 20
Hypertension (Vascular disorders) | 6
Fatigue (General disorders) | 40
Fever w/o neutropenia (General disorders) | 9
Insomnia (Psychiatric disorders) | 3
Weight loss (Investigations) | 12
Dry skin (Skin and subcutaneous tissue disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 29
Nail changes (Skin and subcutaneous tissue disorders) | 6
Pruritus/itching (Skin and subcutaneous tissue disorders) | 5
Rash/desquamation (Skin and subcutaneous tissue disorders) | 12
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 10
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 19
Anorexia (Metabolism and nutrition disorders) | 19
Constipation (Gastrointestinal disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 9
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 20
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 18
Nausea (Gastrointestinal disorders) | 29
Taste disturbance (Nervous system disorders) | 9
Vomiting (Gastrointestinal disorders) | 25
Edema limb (General disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 14
Alkaline phosphatase increased (Investigations) | 11
Alanine aminotransferase increased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 11
Blood bilirubin increased (Investigations) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 5
Creatinine increased (Investigations) | 12
Hyperglycemia (Metabolism and nutrition disorders) | 18
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 8
Dizziness (Nervous system disorders) | 8
Neuropathy-sensory (Nervous system disorders) | 18
Tearing (Eye disorders) | 4
Abdomen, pain (Gastrointestinal disorders) | 3
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 4
Head/headache (Nervous system disorders) | 5
Muscle, pain (Musculoskeletal and connective tissue disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less